CLINICAL TRIAL: NCT01075269
Title: Does Robotic Assistance Significantly Reduce Postoperative Distress and Patient Complaints About Cosmetic Outcomes After Thyroid Surgery? A Preliminary Report.
Brief Title: Postoperative Distress and Cosmetic Outcomes After Open Versus Robotic Thyroidectomy
Acronym: Robot1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korean Association of Endocrine Surgeons (Network)
Responsible Party: Ajou university medical center, department of surgery, Korean Association of Endocrine Surgeons
Other Study IDs: KoreanAES001
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Thyroidectomy; Distress; Surgery
Keywords: robotic thyroidectomy, comparative study, cosmetic result, postoperative neck discomfort, swallowing symptom; Robotic thyroidectomy, cosmetic effect, postoperative distress, surgical outcome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conventional open thyroidectomy group: All patients were told about the operative techniques involved in conventional open and robotic thyroidectomy, and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.
- Robotic thyroidectomy group: All patients were told about the operative techniques involved in conventional open and robotic thyroidectomy, and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.

SUMMARY:
Robotic assistance during thyroid surgery has been utilized clinically in Korea since late 2007. Robotic thyroidectomy has also been validated for surgical management of the thyroid gland. Compared with endoscopic thyroidectomy, the use of a robot in an endoscopic approach via the axilla provides a broader view of the thyroid bed, albeit from a lateral, as opposed to the conventional anterior, perspective. The wrist action of a surgical robot also provides a greater degree of movement than afforded by the use of simple endoscopic instruments, and tremor is eliminated.

Although several reports on operative outcomes of the robotic technique have appeared, no prospective trials comparing the clinical results of robotic with conventional open thyroidectomy have been described. We therefore designed a prospective trial comparing outcomes, including postoperative distress and patient satisfaction, between patients undergoing robotic and conventional open thyroidectomy.

DETAILED DESCRIPTION:
Patient assessment A prospective study addressing perioperative outcomes and postoperative patient discomfort after thyroidectomy was commenced in April 2009 and is currently continuing. All patients were told about the operative techniques involved in conventional open and robotic thyroidectomy, and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent. The study protocol was approved by our Institutional Review Board.

Patients were included if they had (a) a minimally invasive follicular thyroid carcinoma ≤4 cm in diameter, or (b) a papillary thyroid carcinoma ≤2 cm in diameter. Exclusion criteria included (a) previous neck operations; (b) age <21 or >65 years; (c) prior vocal fold paralysis or a history of voice or laryngeal disease requiring therapy; (d) a malignancy with definite extrathyroid invasion, multiple lateral neck node metastasis, perinodal infiltration at a metastatic lymph node, or distant metastasis; and/or (e) a lesion located in the thyroid dorsal area (especially adjacent to the tracheoesophageal groove) caused by possible injury to the trachea, esophagus, or recurrent laryngeal nerve (RLN). The extent of thyroid resection was determined for each patient using American Thyroid Association guidelines. All patients underwent prophylactic ipsilateral central compartment node dissection (CCND; pretracheal, prelaryngeal, and paraesophageal).

Surgical outcomes Surgical outcomes included operating time, intraoperative blood loss, number of retrieved central lymph nodes, length of hospital stay, and postoperative complications. We also assessed the incidence of postoperative seromas and hematomas for at least 3 weeks postoperatively. Operating time was defined as the interval from skin incision to closure. The drainage extent was measured over 24 h, and a drain was removed if drainage was <30 mL in this interval. Study patients were discharged the day after drain removal.

Mobility of the vocal cords was assessed by videostrobolaryngoscopic examination, performed both preoperatively and 1 week and 3 months postoperatively. Vocal cord palsy was defined as permanent when there was no evidence of recovery within 6 months.

Postoperative pain and cosmetic outcomes To evaluate the degree of postoperative pain, all patients were given analgesics on an identical protocol. Patients were asked to grade postoperative pain in the neck and anterior chest as none, very slight, slight, moderate, or severe, 24 h after surgery.

At 1 week and 3 months after surgery, patients were asked (by questionnaire) to evaluate the presence of hyperesthesia and paresthesia in the neck and anterior chest, as well as shoulder discomfort. All patients answered and returned completed questionnaires.

Cosmetic results, including wound appearance and complaints, were evaluated by patients 3 months after surgery using a verbal response scale with five possible responses: extremely satisfied, excellent, acceptable, dissatisfied, and extremely dissatisfied.

Subjective voice and swallowing evaluation We used the Voice Handicap Index-10 (VHI-10), a validated, reliable self-assessment tool that measures patient assessment of voice quality and the effect of voice on quality-of-life, to determine the frequency of voice abnormalities. The VHI-10 consists of 10 questions, responses to each of which are scaled from a minimum of 0 (no voice alteration) to a maximum of 40 (highest voice impairment).

Swallowing difficulties were assessed using the Swallowing Impairment Index (SIS-6), a self-administered, six-item assessment of symptoms related to dysphagia that has been validated for diagnosis of impairment. The scoring of each item on the SIS-6 ranges from a minimum of 0 (no swallowing alteration) to a maximum of 24 (highest swallowing impairment). The SIS-6 score is also excellent for assessing non-voice throat symptoms, including cough, choking, and throat-clearing, all of which occur after thyroidectomy. All patients enrolled in this study completed the VHI-10 and SIS-6 questionnaires before surgery and at 1 week and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* (a) a minimally invasive follicular thyroid carcinoma ≤4 cm in diameter, or
* (b) a papillary thyroid carcinoma ≤2 cm in diameter.

Exclusion Criteria:

* (a) previous neck operations;
* (b) age <21 or >65 years;
* (c) prior vocal fold paralysis or a history of voice or laryngeal disease requiring therapy;
* (d) a malignancy with definite extrathyroid invasion, multiple lateral neck node metastasis, perinodal infiltration at a metastatic lymph node, or distant metastasis; and/or
* (e) a lesion located in the thyroid dorsal area (especially adjacent to the tracheoesophageal groove) caused by possible injury to the trachea, esophagus, or recurrent laryngeal nerve (RLN)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with differentiated thyroid carcinoma who were scheduled to underwent thyroidectomy in Ajou University Medical center (Tertial oncologic center).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Surgical outcomes, postoperative pain and cosmetic outcomes | Postopeative pain: 24 hours after surgery, Cosmetic outcomes: 3 months after surgery
  Surgical outcomes included operating time, intraoperative blood loss, length of hospital stay, and postoperative complications.
  To evaluate the degree of postoperative pain, all patients were given analgesics on an identical protocol. Patients were asked to grade postoperative pain in the neck and anterior chest as none, very slight, slight, moderate, or severe, 24 h after surgery.
  Cosmetic results, including wound appearance and complaints, were evaluated by patients 3 months after surgery using a verbal response scale with five possible responses.

SECONDARY OUTCOMES:
Subjective voice and swallowing evaluation | before surgery and at 1 week and 3 months after surgery.
  We used the Voice Handicap Index-10 (VHI-10), a validated, reliable self-assessment tool that measures patient assessment of voice quality and the effect of voice on quality-of-life, to determine the frequency of voice abnormalities.
  Swallowing difficulties were assessed using the Swallowing Impairment Index (SIS-6), a self-administered, six-item assessment of symptoms related to dysphagia that has been validated for diagnosis of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jandee Lee, MD, Principal Investigator — Korean Association of Endocrine Surgeons
Locations (1):
- Ajou University Medical Center, Department of Surgery, Suwon, South Korea